CLINICAL TRIAL: NCT02115867
Title: Assessment of the Probiotic Symprove as a Dietary Supplement in Patients With Symptomatic Diverticular Disease
Brief Title: Effect of a Probiotic on Diverticular Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12/LO/1695
Record Dates: First submitted 2014-03-20; First posted 2014-04-16 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2014-04

CONDITIONS: Diverticular Disease
Keywords: diverticular disease; diverticulitis; diverticulosis
MeSH Terms: conditions — Diverticular Diseases; Diverticulitis; Diverticulum | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Active Comparator): Probiotic arm Liquid broth
  1 mL/kg every morning for 90 days
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Placebo arm Liquid broth
  1 mL/kg each morning for 90 days
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Symprove probiotic
  Other Names: Symprove probiotic

SUMMARY:
Diverticulitis is an extremely common digestive disease particularly found in the large intestine in elderly patients and develops from diverticulosis. Diverticulosis is characterized by the formation of pouches (diverticula) that bulge to the outside of the colon, through areas of weakness in the colonic wall. Inflammation (diverticulitis) results if one of these diverticula becomes infected and / or obstructed. It is commonly accompanied by obvious or microscopic perforation, ranging in severity from a single, mild, acute attack of diverticulitis to more severe attacks characterized by abscess formation, occasionally resulting in chronic complications such as obstruction and fistula formation. After an episode of diverticulitis many patients develop changes in bowel openings, from diarrhoea and constipation, and many patients have abdominal pain and a symptom complex that resembles Irritable Bowel Syndrome (IBS).

According to available guidelines, treatment of symptomatic, but uncomplicated, diverticular disease aims to reduce the frequency and severity of diverticular related symptoms (abdominal pain, bloating, alterations in bowel habit) and to prevent complications. Different agents have been proposed, such as bulking agents, antispasmodics, and nonabsorbed topical antibiotics, 5amino acid preparations but these measures are unproven or controversial. It is thought that intestinal bacteria may play a significant role in the symptoms of post-diverticulitis.

The investigators have recently shown that a probiotic (Symprove) reduced the symptoms of IBS significantly in comparison with a placebo in a double-blind randomized trial and without side effects (paper in preparation). Because the symptoms in IBS and post-diverticulitis are so similar the investigators propose a double-blind placebo controlled trial of Symprove in patients with problematic diverticulitis. Patients will be recruited from a dedicated diverticulitis clinic using standard exclusion criteria. This is a 90 day symptom based trial using accepted outcome measures. If successful the results will have widespread implications for treatment of diverticular disease.

DETAILED DESCRIPTION:
The patients for this study will be recruited from the diverticular disease clinic at King's College Hospital. The clinic is the first and the largest specialist diverticular clinic in the UK and attracts referrals directly from GP's, internal referrals from gastroenterology, in and outpatients and increasingly from Gastroenterology and Colorectal Surgery clinics in the South East of England. Eligible patients who meet fulfill the entry criteria will be invited to participate. They will receive a patient information sheet, which they take home with them for reading. They will then be seen again (usually within 2 weeks, or after any confirmatory tests have been completed) to discuss any questions that they may have and for a decision for inclusion into the trial.

Each will undergo a full blood count and conventional biochemistry and they will provide a stool sample for assessment of intestinal inflammation by a calprotectin estimation. They will also complete a baseline symptoms-based questionnaire. They will then be randomized to treatments A or B, both investigator and patient will be unaware of whether it is the active treatment (Symprove) or placebo. Each patient will complete the symptom-based questionnaire every 30 days while on on the 90 day treatment (Day 30, Day 60, and Day 90). The primary outcome measure will be a change in symptoms score from Day 0 to Day 90.

Also every 30 days while on treatment, stool tests will be repeated for faecal calprotectin. An additional sample will be frozen for eventual microbiota assessment. The secondary outcome measure will be change in the faecal microbiota between Day 0 and Day 90.

Patients will be seen in clinic 30 days after cessation of the trial (Day 120), at which time those patients on placebo will be offered a 90 day free treatment with the active ingredient if they so wish.

ELIGIBILITY:
Inclusion Criteria:

* Have a documented episode of diverticulitis as assesses clinically, on CT scans and a raised serological markers of inflammation
* Have problematic symptoms associated with established diverticular disease, post a diverticulitis episode
* Aged over 20 years
* Are on no treatment or have been on stabile medication for at least 6 weeks for diverticular disease
* Willing and able to provide a written informed consent.

Exclusion Criteria:

* Aged less than 20 years
* Severe disease (ongoing severe active diverticulitis) as defined by hemoglobin < 8.0 g/dl, white blood cell count, >20,000 cells/mm3, temperature >38.5°C, serum albumin < 25 g/dl
* Surgical diverticular complications such as rectovaginal or bladder fistula, abscess, etc.
* Severe respiratory, cardiovascular, neurological, psychiatric, rheumatological, other gastrointestinal, etc. diseases
* Undergone major intestinal resections
* Patients with malignancy
* On NSAIDs
* Pregnancy or actively seeking pregnancy
* History of intolerance or allergy to probiotics
* Current drug or alcohol dependence syndrome
* Patients unable to consent for themselves
* Patients with severe learning difficulties

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2013-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in symptoms assessment score | 90 days
  The primary outcome in this study is the postulated improvement in symptom severity scores over the 90 day treatment period. There is no generally approved or validated symptom severity scoring system for patients with diverticular disease. In view of the fact that the symptoms (and possible the cause of symptoms) of post-diverticulitis is almost identical to that of IBS we propose to use this scoring system and we have added a separate additional pain score outcome as this is the principal symptoms that diverticulitis patients experience. In addition to the symptoms based assessment, patients will complete an SF-8 questionnaire. Both questionnaires will be completed prior to treatment initiation (Day 0) and again at the end of treatment (Day 90). The change from baseline symptoms score to symptoms score at Day 90 will be the primary outcome measurement.

SECONDARY OUTCOMES:
Change in faecal microbiota | 90 days
  Patients will submit a stool sample prior to treatment initiation and every 30 days after initiating treatment for assessment of faecal microbiota (Day 30, 60, and 90). The secondary outcome measure for the study will be change in faecal microbiota between Day 0 and Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Ingvar Bjarnason, MD, MSc, Principal Investigator — King's College Hospital NHS Trust; Savvas Papagrigoriadis, MD, MSc, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No